CLINICAL TRIAL: NCT00698477
Title: Study of the Effect of Chemotherapy on Methylation Patterns in Breast Tumor Tissue and Paired Plasma Samples and Correlation With Clinical Response and Outcomes
Brief Title: Chemotherapy on Methylation Patterns in Breast Tumor Tissue Correlating With Clinical Response and Outcomes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Other Study IDs: BR04/19/07
Record Dates: First submitted 2008-06-15; First posted 2008-06-17 (Estimated); Last update posted 2008-06-17 (Estimated); Status verified 2008-06

CONDITIONS: Breast Tumor Tissue

SUMMARY:
Primary Objectives

1. To identify hypermethylated genes in paired pretreatment breast tumor tissue and plasma samples from locally advanced and metastatic breast cancer patients using a known gene panel which includes APC1, Cyclin D2, RARB, RASSF1A, Twist, Hin1 and GSTP1.

   Rationale: We and others have determined the optimal panel of genes that are able to detect free DNA in plasma and serum. We will determine if the same panel of genes is effective for detecting tumor DNA in the plasma of locally advanced and metastatic breast cancer patients. Further, to determine if the methylation profile of the plasma DNA for these genes is the same or different from the primary tumor at presentation, we will analyze the primary tumor DNA from fresh frozen samples.
2. To identify methylation pattern changes in the same subset of patients' plasma samples at 24 hours after completion of cycle 1 of chemotherapy and within 24 hours before cycle 2.

Rationale: The optimal timing of sampling for methylation analysis that is reflective of the tumors response to chemotherapy is not known. How soon methylation changes are observed, whether they are high within 24 hours, as that tumor responds to chemotherapy, or whether changes can be observed only some time after one cycle of chemotherapy will be studied. (3) To also identify methylation pattern changes in breast tumor tissue after one cycle of chemotherapy.

Rationale: To look for a correlation with plasma methylation patterns

Secondary Objectives

(1) To correlate our observed patterns of methylation pre- and post-treatment with clinical parameters such as clinical and/or radiological response and patient outcome.

DETAILED DESCRIPTION:
In advanced breast cancer, it is often difficult to predict which patients will respond favorably to systemic therapy to decide on treatment duration or options while minimizing exposure to toxic effects. Our goal is to examine using locally advanced and metastatic breast cancer tumor tissue and plasma, the methylation profile patterns pre- and post chemotherapy of a panel of biomarkers most commonly expressed in breast cancer and correlate them with tumor response and patient outcome.

Our hypothesis is that DNA methylation pattern changes at baseline and early into a course of systemic therapy can predict disease response or progression as well as survival. In the long term, this could prove clinically useful in limiting exposure to ineffective regimens and allowing earlier identification of more effective systemic therapy.

Core biopsies of breast tumor tissue are taken at baseline and after cycle 1 of docetaxel/ketoconazole. Plasma samples are drawn at baseline, 24 hours after cycle 1 chemotherapy and 24 hours before cycle 2. Thirty patients' specimens (60 core biopsies and 90 plasma samples) will be utilized. Quantitative multiplex methylation-specific PCR will be used for analyses of several tumor suppressor genes including APC1, Cyclin D2, RARB, RASSF1A, Twist, Hin1 and GSTP1. From this data, we will identify a preliminary gene panel associated with breast cancer which undergoes the most changes in methylation following systemic therapy. Thirty paraffin-embedded healthy tissue samples from mastectomy specimens and blood samples from unaffected individuals will serve as normal controls.

This preliminary study can be used to determine the clinical utility of DNA methylation in breast tumor tissue and plasma as a predictive marker for response to chemotherapy and a prognostic marker for patient outcome. If a relationship is found, we can then further study if the change in methylation pattern has clinical utility in influencing therapeutic decision-making which may be further expanded to the adjuvant setting..

ELIGIBILITY:
Inclusion Criteria:

We are not actively recruiting breast cancer patients but using stored biospy and plasma samples collected in the stated Clinical Trial (Phase II study of docetaxel combined with ketoconazole in the first-line treatment of locally advanced or metastatic breast cancer patients with measurable primary breast tumor) which was already IRB-approved

For the normal controls, inclusion criteria are:

1. Any female adult patient above 21
2. No current or past history of underlying malignancies

Exclusion Criteria:

For normal controls, exclusion criteria are:

(1) Past or current history of malignancies

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2007-10

CONTACTS AND LOCATIONS:
Overall Officials: Sing Huang Tan, MBBS, MRCP, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

REFERENCES:
- [Background] Fackler MJ, McVeigh M, Mehrotra J, Blum MA, Lange J, Lapides A, Garrett E, Argani P, Sukumar S. Quantitative multiplex methylation-specific PCR assay for the detection of promoter hypermethylation in multiple genes in breast cancer. Cancer Res. 2004 Jul 1;64(13):4442-52. doi: 10.1158/0008-5472.CAN-03-3341. PMID 15231653
- [Background] Swift-Scanlan T, Blackford A, Argani P, Sukumar S, Fackler MJ. Two-color quantitative multiplex methylation-specific PCR. Biotechniques. 2006 Feb;40(2):210-9. doi: 10.2144/000112097. PMID 16526411